CLINICAL TRIAL: NCT07220811
Title: Phase 2b Randomized, Double-Blind, Placebo-Controlled Study of RPT904 as Monotherapy in Participants With IgE-Mediated Food Allergy
Brief Title: Phase 2b Study of RPT904 as Monotherapy in Participants With IgE-Mediated Food Allergy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RAPT Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RPT904-01
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Ig-E Mediated Food Allergy
Keywords: Ig-E Mediated food allergy; peanut allergy; milk allergy; egg allergy; cashew allergy; walnut allergy; RPT904; placebo; double-blind placebo-controlled food challenge (DBPCFC); ozureprubart; JYB1904
MeSH Terms: conditions — Peanut Hypersensitivity; Milk Hypersensitivity; Egg Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RPT904 (Q8W) (Experimental): RPT904 every 8 weeks. The dose levels of RPT904 (150 mg, 300 mg, and 600 mg) within the Q8W cohort will be assigned based on participant weight and baseline total IgE level.
  RPT904 subcutaneous injection every 8 weeks with a loading dose at Week 2 (Part 1: 24 weeks; Part 2: 24 weeks); matching placebo at intervening visits to maintain blinding.
  Interventions: Drug: RPT904; Other: Placebo
- RPT904 (Q12W) (Experimental): RPT904 every 12 weeks. The dose levels of RPT904 (150 mg, 300 mg, and 600 mg) will be assigned based on participant weight and baseline total IgE level.
  RPT904 subcutaneous injection every 12 weeks with a loading dose at Week 2 (Part 1: 24 weeks; Part 2: 24 weeks); matching placebo at intervening visits to maintain blinding.
  Interventions: Drug: RPT904; Other: Placebo
- Placebo (Placebo Comparator): Placebo subcutaneous injection on schedules matching both the Q8W and Q12W arms in Part 1 (24 weeks); RPT904 every 8 or 12 weeks with a loading dose at Week 26 on schedules matching both the Q8W and Q12W arms Part 2 (24 weeks), with matching placebo at intervening visits to maintain blinding.
  Interventions: Drug: RPT904; Other: Placebo

INTERVENTIONS:
Drug: RPT904 — Subcutaneous injection once every 8 weeks
  Other Names: ozureprubart; JYB1904
  Arms: RPT904 (Q8W)
Drug: RPT904 — Subcutaneous injection once every 12 weeks
  Other Names: ozureprubart; JYB1904
  Arms: RPT904 (Q12W)
Other: Placebo — Subcutaneous injection at the intervening dosing visits
  Arms: RPT904 (Q12W); RPT904 (Q8W)
Drug: RPT904 — Subcutaneous injection once every 8 weeks (Part 2)
  Other Names: ozureprubart; JYB1904
  Arms: Placebo
Drug: RPT904 — Subcutaneous injection once every 12 weeks (Part 2)
  Other Names: ozureprubart; JYB1904
  Arms: Placebo
Other: Placebo — Subcutaneous injection on schedules matching both the Q8W and Q12W arms (Part 1). Subcutaneous injection at the intervening dosing visits (Part 2)
  Arms: Placebo

SUMMARY:
Phase 2b Study of RPT904 as Monotherapy in Participants With IgE-Mediated Food Allergy: This is a Phase 2b randomized, double-blind, placebo-controlled clinical trial evaluating RPT904, a next-generation anti-IgE monoclonal antibody, in people with food allergy. RPT904 is a long-acting antibody that may allow for dosing every 8 to 12 weeks. Approximately 100 participants between the ages of 12 and 55 with documented allergy to at least one of the following foods: peanut, milk, egg, cashew, or walnut will be enrolled. In Part 1 (24 weeks), participants will be randomly assigned to receive RPT904 every 8 or 12 weeks (plus a loading dose at Week 2), or placebo. In Part 2 (24 weeks), participants who received RPT904 will continue on their assigned dosing schedule, and those who previously received placebo will be re-randomized to receive RPT904 either every 8 or 12 weeks (plus a loading dose at Week 26). All participants will attend study visits approximately every 2-6 weeks throughout both Part 1 and Part 2 to maintain blinding, regardless of treatment group or dosing frequency. The study is being conducted at multiple sites. The primary goal is to assess whether RPT904 helps participants tolerate higher amounts of a food allergen without dose-limiting allergic symptoms during a food challenge. The study will also monitor the safety and side effects of RPT904 over time. Each participant is expected to be in the study for about 68 to 74 weeks, including screening, treatment, and follow-up.

DETAILED DESCRIPTION:
Phase 2b Randomized, Double-Blind, Placebo-Controlled Study of RPT904 as Monotherapy in Participants With IgE-Mediated Food Allergy

ELIGIBILITY:
Key Inclusion Criteria:

* Participant and/or parent/legal guardian must be able to understand and provide informed consent and/or assent, as applicable.
* Male or female, 12 to less than 56 years of age at screening.
* Allergic to at least 1 of the following foods: peanut, milk, egg, cashew, or walnut, as confirmed by the following criteria:
* a. For participants aged 12 to <18 years:
* i. Allergic to peanut: participant must meet all criteria below:
* 1. Positive SPT (≥4 mm wheal greater than saline control) to peanut.
* 2. Positive peanut IgE (≥6 kUA/L) at screening or within 3 months of screening.
* 3. Positive blinded oral food challenge (OFC) to peanut during the screening DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤100 mg (ie, cumulative dose of ≤144 mg) of peanut protein.
* ii. Allergic to milk or egg: unable to tolerate both cooked and uncooked forms:
* 1. Positive SPT (≥4 mm wheal greater than saline control) to the specific food.
* 2. Positive food-specific IgE (≥6 kUA/L) at screening or within 3 months of screening.
* 3. Positive blinded OFC to the specific food during the screening DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤300 mg (ie, cumulative dose of ≤444 mg) of food protein.
* iii. Allergic to cashew: participant must meet all criteria below:
* 1. Positive SPT (≥4 mm wheal greater than saline control) to cashew. OR
* 2. Positive cashew IgE (≥6 kUA/L) at screening or within 3 months of screening. AND
* 3. Positive blinded OFC to cashew during the screening DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤100 mg (ie, cumulative dose of ≤144 mg) of cashew protein.
* iv. Allergic to walnut: participant must meet all criteria below:
* 1. Positive SPT (≥4 mm wheal greater than saline control) to walnut. OR
* 2. Positive walnut IgE (≥6 kUA/L) at screening or within 3 months of screening AND
* 3. Positive blinded OFC to walnut during the screening DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤300 mg (ie, cumulative dose of ≤444 mg) of walnut protein.
* b. For participants aged 18 to <56 years:
* i. Allergic to peanut or cashew: participant must meet all of the following criteria:
* 1. Positive SPT (≥3 mm wheal greater than saline control) to peanut or cashew.
* 2. Positive peanut or cashew IgE (≥0.35 kUA/L) at screening or within 3 months of screening.
* 3. Positive blinded OFC to peanut or cashew during the screening DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤100 mg (ie, cumulative dose of ≤144 mg) of peanut or cashew protein.
* ii. Allergic to milk or egg: participant must meet all of the following criteria:
* 1. Positive SPT (≥3 mm wheal greater than saline control) to the specific food.
* 2. Positive food-specific IgE (≥0.35 kUA/L) at screening or within 3 months of screening.
* 3. Positive blinded OFC to the specific food during the screening DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤300 mg (ie, cumulative dose of ≤444 mg) of food protein.
* iii. Allergic to walnut: participant must meet all of the following criteria:
* 1. Positive SPT (≥3 mm wheal greater than saline control) to walnut.
* 2. Positive walnut IgE (≥0.35 kUA/L) at screening or within 3 months of screening.
* 3. Positive blinded OFC to walnut during the screening DBPCFC, defined as experiencing dose-limiting symptoms at a single dose of ≤300 mg (ie cumulative dose of ≤444 mg) of walnut protein.
* With body weight (as measured at screening) and total serum IgE level (as measured within 3 months of screening) suitable for RPT904 dosing (per RPT904 dosing table).
* Female Participants:
* 1. Must not be pregnant or breastfeeding.
* 2. Women of non-childbearing potential (e.g., surgically sterile or postmenopausal) are eligible.
* 3. Women of childbearing potential must have a negative pregnancy test before starting study treatment, agree to use a protocol-defined method of contraception during the study and for at least 16 months after the last dose, and must not donate eggs or undergo egg retrieval during this period.
* Male Participants:
* 1. Must agree to either remain abstinent from heterosexual intercourse (if that is their usual lifestyle) or use protocol-defined contraception during the study and for 16 months after the last dose.
* 2. Must not donate semen or participate in sperm banking during this time, and if they have a female partner of childbearing potential, she should also use effective contraception.

Exclusion Criteria:

* Clinically significant lab abnormalities at screening.
* Sensitivity or suspected/known allergy to any component of the active or placebo OFC material (excluding the test allergens peanut, milk, egg, walnut, and cashew being tested), or drugs related to RPT904 (eg, monoclonal antibodies, polyclonal gamma globulin).
* Uncontrolled or severe asthma/wheezing at screening.
* Current use of oral, IM, or IV corticosteroids, tricyclic antidepressants, or β-blockers (oral or topical).
* Past or current immunotherapy to any study foods within 6 months of screening.
* Treatment with immunomodulatory therapy within 6 months of screening.
* Currently in the "build-up phase" of inhalant allergen immunotherapy (i.e., not yet on maintenance). Note: individuals on stable maintenance dosing may be eligible.
* Past or current medical problems (eg, severe latex allergy), chronic diseases (other than asthma/wheezing, atopic dermatitis, or rhinitis) requiring therapy (eg, heart disease, diabetes), abnormal physical findings or lab results not listed above that, in the Principal Investigator's opinion, may increase study related risks, hinder protocol compliance, or impact data quality or interpretation .

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To compare the ability to consume a food without dose-limiting symptoms during a DBPCFC at the end of Part 1 after treatment with either RPT904 or placebo | Approximately 24 weeks
  Proportion of participants who consumed a single dose of ≥600 mg (ie, a cumulative dose of ≥1044 mg) of peanut or cashew protein, or a single dose of ≥1000 mg (ie, a cumulative dose of ≥2044 mg) of milk, egg, or walnut protein without dose-limiting symptoms at Part 1 DBPCFC

SECONDARY OUTCOMES:
To evaluate safety during treatment with either RPT904 or placebo | Approximately 48 weeks
  Frequency of treatment-emergent adverse events (TEAEs) related to study therapy regimen

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Arkansas Children's, Little Rock, Arkansas
  - Asthma & Allergy Associates, P.C., Colorado Springs, Colorado
  - Children's Healthcare of Atlanta - Center for Advanced Pediatrics, Atlanta, Georgia
  - Clinical Research Institute, Inc, Minneapolis, Minnesota
  - Northwell Health, Great Neck, New York
- Children's Hospital at Westmead, Westmead, New South Wales, Australia
- Canada (2):
  - Halton Pediatric Allergy, Burlington, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No